CLINICAL TRIAL: NCT06549543
Title: Additional Effect of High-Intensity Laser Therapy Over Conventional Physiotherapy Related to Pain and Function in Patients With Knee Osteoarthritis: A Randomized, Double-Blind, Placebo-Controlled, 12-Week Follow-up Study
Brief Title: High-Intensity Laser Therapy: Effectiveness on Knee Osteoarthritis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Selen Özgözen, Clinical Doctor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KA22/129
Record Dates: First submitted 2024-08-02; First posted 2024-08-12 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Osteoarthritis, Knee
Keywords: high-intensity laser; rehabilitation; pain; osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Osteoarthritis | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: patients were assigned into two groups. Both groups received conventional physiotherapy and exercise therapy. Group 1 was the experimental group, and group 2 was the control group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Both the participants, investigators and outcomes assessors were blinded throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-Intensity Laser Therapy (Experimental): This group (n = 21) received transcutaneous electrical nerve stimulation (TENS), hotpack (HP), exercises, and high-intensity laser therapy (HILT) for 10 consecutive sessions.
  Interventions: Other: High Intensity Laser Therapy; Other: Transcutaneous Electrical Nerve Stimulation; Other: Hotpacks
- Control (Sham Comparator): This group (n = 22) received TENS, HP, exercises, and placebo HILT for 10 consecutive sessions.
  Interventions: Other: Transcutaneous Electrical Nerve Stimulation; Other: Hotpacks; Other: SHAM - High Intensity Laser Therapy

INTERVENTIONS:
Other: High Intensity Laser Therapy — HILT is applied per session, with a maximum of 10.0 W, a mean of 5.7 W, a dose of 99 J/cm², and a total energy flux of 2079 J were applied over 6 minutes and 5 seconds on a 21 cm² field on the medial aspect of the knee joint.
  Arms: High-Intensity Laser Therapy
Other: Transcutaneous Electrical Nerve Stimulation — TENS is an analgesic modality of physical therapy
Other: Hotpacks — Hotpacks is a thermoanalgesia modality of physical therapy
Other: SHAM - High Intensity Laser Therapy — for control group, sham HILT was applied, with lights on but no laser beam
  Arms: Control

SUMMARY:
The aim of this prospective, randomized, double-blinded study is to investigate the additional benefits of high-intensity laser therapy (HILT) over conventional physiotherapy, related to pain and function, in patients with knee osteoarthritis (KOA).

DETAILED DESCRIPTION:
The study was performed in Baskent University Physical Therapy and Rehabilitation Unit. 43 patients of both sexes, who were diagnosed clinical and radiographic knee osteoarthritis, with Kellgren Lawrence Grade 2 and 3, were randomly assigned in two groups. Group 1 (n = 21) received TENS, HP, exercises (EX), and High-Intensity Laser Therapy (HILT; Nd:yag laser, 10W). Group 2 (n = 22) received the same interventions but placebo HILT. All interventions were applied for 10 sessions. The Visual Analog Scale (VAS), Western Ontario & McMaster Universities Osteoarthritis Questionnaire (WOMAC), and Lequesne Algofunctional Index (LAI) were performed before, after, and at 12-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* both sexes and age between 40 and 65;
* pain at least 3 months on single or both knees
* diagnosed as KOA with Kellgren Lawrence (KL) Grade 2 or 3 KOA on weight-bearing anteroposterior X-ray images
* normal serum acute phase reactants and uric acid levels
* had no major effusion in the joint.

Exclusion Criteria:

* therapeutic joint injection in the last 6 months
* physical therapy and/or HILT in the last 3 months
* any surgical invention for the knee joint
* malignancy in the last 5 years.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
The Visual Analog Scale (VAS) | 12 weeks
  The VAS was assessed before treatment, at the end of 10 sessions, and at the 12 week follow-up. Min score was 0 and max score was 100. Higher scores on the VAS indicate greater pain.

SECONDARY OUTCOMES:
Western Ontario & McMaster Universities Osteoarthritis Questionnaire (WOMAC) | 12 weeks
  The WOMAC was assessed before treatment, at the end of 10 sessions, and at the 12 week follow-up. Higher scores on the WOMAC indicate poorer functional capacity and greater pain and stiffness.
Lequesne Algofunctional Index (LAI) | 12 weeks
  The LAI was assessed before treatment, at the end of 10 sessions, and at the 12 week follow-up. Higher scores on the LAI indicate poorer functional capacity and greater pain and stiffness.

CONTACTS AND LOCATIONS:
Locations (1):
- Başkent University Faculty of Medicine, Yüreğir, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akaltun MS, Altindag O, Turan N, Gursoy S, Gur A. Efficacy of high intensity laser therapy in knee osteoarthritis: a double-blind controlled randomized study. Clin Rheumatol. 2021 May;40(5):1989-1995. doi: 10.1007/s10067-020-05469-7. Epub 2020 Oct 19. PMID 33074393
- [Background] Ekici B, Ordahan B. Evaluation of the effect of high-intensity laser therapy (HILT) on function, muscle strength, range of motion, pain level, and femoral cartilage thickness in knee osteoarthritis: randomized controlled study. Lasers Med Sci. 2023 Sep 25;38(1):218. doi: 10.1007/s10103-023-03887-y. PMID 37743421
- [Background] Hardie EM, Carlson CS, Richardson DC. Effect of Nd:YAG laser energy on articular cartilage healing in the dog. Lasers Surg Med. 1989;9(6):595-601. doi: 10.1002/lsm.1900090610. PMID 2601554
- [Background] Ahmad MA, A Hamid MS, Yusof A. Effects of low-level and high-intensity laser therapy as adjunctive to rehabilitation exercise on pain, stiffness and function in knee osteoarthritis: a systematic review and meta-analysis. Physiotherapy. 2022 Mar;114:85-95. doi: 10.1016/j.physio.2021.03.011. Epub 2021 Mar 26. PMID 34654554